CLINICAL TRIAL: NCT02828722
Title: Proof of Concept Trial to Confirm That the Recovery of Patients Treated in the Intensive Care Unit Requiring Mechanical Ventilation is Beneficially Affected by the Environmental Simulation of Daytime and Night Time Alternation as Well as by the Nutrition Protocol Corresponding to the Daily Rhythm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Achros Health Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACHROS CRC-003
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Critical Illness; Mechanical Ventilation
Keywords: Circadian rhythm; Critical Illness; Mechanical ventilation; Environmental modulation
MeSH Terms: conditions — Critical Illness | interventions — Noise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Controlled light, noise and nutrition (Experimental): Simultaneously with the standard treatment performed at the clinical trial site environmental simulation of night time and daytime alternation as well as the nutrition protocol corresponding to the daily rhythm will be applied.
  Interventions: Other: Controlled light and noise; Other: Controlled nutrition
- Controlled light and noise (Experimental): Simultaneously with the standard treatment performed at the clinical trial site environmental simulation of night time and daytime alternation as well as the continuous nutrition (in accordance with the clinical trial site's standard practice) will be applied.
  Interventions: Other: Controlled light and noise
- Control (No Intervention): The treatment of the study subject will be performed based on the clinical trial site's standard practice without environmental simulation or changes in the nutrition protocol.

INTERVENTIONS:
Other: Controlled light and noise — Purpose: The day-night ratio of the environmental illumination (limit 8 lux) and that of the noise level (limit 20 dBA) must correspond to the necessary value required by a healthy human body as defined by the National Sleep Foundation (USA).
  Implementation: Simulation of the daytime period is performed with blue predominant artificial light with colour temperature between 5500 and 8000 K with lux values of 1000-1200 measured at the head of the patient. Simulation of the nighttime period is performed with a sleeping mask and earplugs.
  Other Names: Environmental simulation of the daytime and night time alternation
  Arms: Controlled light and noise; Controlled light, noise and nutrition
Other: Controlled nutrition — In compliance with the standard daily nutrition protocol, nutrition is carried out only during daytime both in case of enteral and parenteral feeding in accordance with European Society for Clinical Nutrition and Metabolism 2016 guidelines.
  Nutritional regimen should be stopped for 8 hours/24 at night (non-nutritional period may be depending on the work schedule of the actual ICU) , even if the daily energy/protein target is not reached.
  Other Names: Nutrition protocol that is in accordance with the daily rhythm
  Arms: Controlled light, noise and nutrition

SUMMARY:
The purpose of this study is to determine whether the environmental simulation of daytime and night time alternation as well as by the nutrition protocol corresponding to the daily rhythm are beneficially affect the recovery of patients treated in the Intensive Care Unit (ICU) requiring mechanical ventilation.

DETAILED DESCRIPTION:
The homeostasis of human body is significantly disturbed when organs' work-relax periods are not harmonized. Intensive Care Unit (ICU) patient's circadian rhythm is almost inevitably upset as a result of their disease and/or medical intervention. There are numerous animal studies prove that circadian rhythm and periodic dynamics are directly related to healing time and hence, mortality rate. Although, one of the main messengers of circadian synchronization is melatonin, it is overridden by temperature, and a number of other factors from e.g. the digestive tract. If the circadian rhythm is disturbed, the function of different organ systems becomes desynchronized and chaotic.

ICU environment and patient-care activities brings major drawbacks as well mainly by necessary presence of noise and light. It has been shown that ICU settings have an impact on patients' sleep, which can easily lead to delirium and circadian disruption. There are significant data showing strong correlation between delirium and ICU length of stay/ mortality.

The focus of this study is the environmental modulation at the ICU with controlled light, noise and nutrition conditions. Controlled light conditions are created with artificial light during daytime and sleeping mask during night time. Earplugs are used during night time for controlled noise conditions. Nutrition is carried out only during daytime both in case of enteral and parenteral feeding.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Requiring treatment at the intensive care unit including mechanical ventilation
* Admission at the intensive care unit was done within 24 hours before randomization
* Written and signed patient information sheet and informed consent form obtained by the study participant or by his/her legal representative

Exclusion Criteria:

* Traumatic brain injury
* Multiple trauma
* Severe damage of the eye/optic nerve
* Blindness
* Post CPR
* Unlikely to survive 24 hours
* Involvement of the central nervous system (trauma, bleeding, infection, ischemia, etc.)
* Intracranial space occupying process
* Increased intracranial pressure
* Narcolepsy
* Huntington's disease
* Hypothermia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change of the Multiple Organ Dysfunction Score value (delta MODS) from baseline to the end of the study treatment | Over the ICU treatment period but no more than 10 days
  The primary efficacy endpoint is the change in MODS scale from baseline to the end of the study treatment period, i.e. deltaMODS. Since the length of ICU stay may be different for subjects, the MODS rate of change per day (deltaMODS/day) will be the primary measure to characterize the treatment effect.

SECONDARY OUTCOMES:
Change of the MODS value (delta MODS) between worst and last score during the study treatment | Over the ICU treatment period but no more than 10 days
  Change of the MODS value between worst and last score over the ICU treatment period but no longer than 10 days.
Number of participants with gastric retention | over the ICU treatment period but no more than 10 days
  Number of participants with at least 250ml gastric retention at least one time
Number of participants with delirium | over the ICU treatment period but no more than 10 days
  Number of participants with at least one evaluated Intensive Care Delirium Screening Checklist (ICDSC) score between 4-8

OTHER OUTCOMES:
Change of the acute physiology and chronic health evaluation II (APACHE II) score from baseline to the end of the study treatment | during study participation but but no more than 10 days
Change of the Sequential Organ Failure Assessment (SOFA) score from baseline to the end of the study treatment | during study participation but but no more than 10 days
Change of the Simplified Acute Physiology II score (SAPS II) score from baseline to the end of the study treatment | during study participation but but no more than 10 days
average daily dose of sedatives | during study participation but but no more than 10 days
length of ICU treatment from admission to discharge in days | during study participation but no more than 99 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged Faculty of Medicine, Department of Anaesthesiology and Intensive Therapy, Szeged, Hungary